CLINICAL TRIAL: NCT03028844
Title: The Effect of a Musical Intervention on Stress Response to Venepuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Dr. Gene Dempsey, Prof, University College Cork
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ED/01/16UCC
Record Dates: First submitted 2017-01-09; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pain; Stress, Physiological
Keywords: Neonate; preterm; pain; music; EEG; venepuncture
MeSH Terms: conditions — Pain; Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose alone (No Intervention): These infants will receive an oral sucrose solution ("Sweetease") only prior to venepuncture
- Music intervention plus sucrose (Experimental): These infants will receive both oral sucrose solution and music therapy prior to venepuncture.
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — The musical intervention will be played for ten minutes prior to venepuncture
  Arms: Music intervention plus sucrose

SUMMARY:
Randomised Crossover Trial in Preterm Infants less than 32 weeks to assess Music therapy and sucrose versus sucrose on stress

DETAILED DESCRIPTION:
The purpose of this study is to assess whether the use of music therapy as a non-pharmacological intervention around the time of venepuncture significantly decreases the stress response of a stable preterm neonate, as measured by salivary cortisol levels .

The secondary aim of this study is to analyse the effect of music therapy on the EEG, and vital signs of the stable preterm neonate.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at less than 32 weeks gestational age (from 23+0 weeks' up to and including 31+6 weeks' gestational age)
* Infants must now be >32 weeks corrected gestational age
* Infants who are medically stable and due to have routine venepuncture as part of their management plan

Exclusion Criteria:

* Inability to obtain informed consent from parent
* Infants with known hearing impairment
* Infants receiving sedative medications
* Any evidence of dysfunction of the hypothalamic-pituitary-adrenal axis
* Infants with congenital abnormalities
* Infants with known EEG abnormalities

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol levels | BASELINE, 20 mins and 4 hours
  Change in salivary cortisol levels between Baseline, 20 minutes and 4 hours

SECONDARY OUTCOMES:
Premature Infant Pain Profile (PIPP) score | immediate
  Alteration in pain as measured by Premature Infant Pain Profile (PIPP) score
Changes in physiological parameters - Heart rate | 10 mins before venepuncture and 10 mins after
  Increase in heart rate
Changes in physiological parameters - respiration rate | 10 mins before venepuncture and 10 mins after
  Increase in respiration rate
Changes in physiological parameters - oxygen saturation | 10 mins before venepuncture and 10 mins after
  Decrease in oxygen saturation
Changes in physiological parameters - EEG | 10 mins before venepuncture and 10 mins after
  Altered EEG amplitude and Frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Maternity Hospital, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No